CLINICAL TRIAL: NCT07069777
Title: Muscle Quality and Subcutaneous Adipose Tissue in the Rectus Femoris and Rectus Abdominis Muscles: Ultrasound Evaluation and Functional Correlation in Older Adults
Status: Not yet recruiting | Type: Observational
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, Luis Polo Ferrero, Associate Professor of Physical Therapy at the University of Salamanca, University of Salamanca
Other Study IDs: USalamancaOSRFRA
Record Dates: First submitted 2025-07-07; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-05

CONDITIONS: Ultrasound; Sarcopenia; Obesity
Keywords: ultrasound; obesity; sarcopenia; muscle quality; active aging
MeSH Terms: conditions — Sarcopenia; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (4):
- Obesity with low strenght: BMI >30 and/or waist circumference of 88 cm or more and grip strength <16 kg.
- Obesity with normal strength: BMI >30 and/or waist circumference of 88 cm or more and grip strength >16 kg.
- Non-obesity with normal strength.: BMI <30 and/or waist circumference less than 88 cm and grip strength >16 kg.
- Non-obesity with low strength.: BMI <30 and/or waist circumference less than 88 cm and grip strength <16 kg.

SUMMARY:
The goal of this observational, cross-sectional study is to examine the relationship between body composition and muscle quality in women over the afe of 65. The main question it aims to answer is:

How are ultrasound-based measurements of muscle and fat tissue related to functional performance in older women?

DETAILED DESCRIPTION:
In this observational and cross-sectional study, researchers will use ultrasound imaging and physical performance tests to evaluate muscle thickness, subcutaneous fat thickness, abdominal circumference, handgrip strength, and functional performance. These measurements will help identify muscle and fat distribution profiles associated with higher functional risk in older adults.

This study aims to contribute to the understanding of sarcopenic obesity and muscle quality in aging, with the ultimate goal of improving preventive physiotherapy strategies and promoting healthy aging.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 65 years and living in the community.
* Female sex.
* Enrolled as a participant in PReGe program.

Exclusion Criteria:

* Recent surgery (<6 months) involving the abdomen or lower extremities.
* Presence of methal prostheses or implants in the thigh or abdoinal region.
* Diagnosed neuromuscular disease (e.g., myopathies, advanced Parkinson's disease.)
* Musculoskeletal disorders that impair basic mobility or prevent functional testing.
* Acute illness or clinical decompensation at the time of assessment.
* Unintentional weight loss > 5 kg within the past month (suggestive of cachexia risk).
* Presence of active abdominal hernias or severe diastasis recti.

Min Age: 65 Years | Sex: Female
Age Groups: Older Adult
Study Population: Community-dwelling women aged 65 years and older participating in the PReGe (research on active aging with preventive physiotherapy) project. The population is generally independent in activities of daily living and not institutionalized
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Ultrasound Assessment of the Rectus Femoris Muscle | At a single assessment visit
  The rectus femoris muscle was assessed using B-mode ultrasound imaging, following SARCUS group recommendations. Participants were positioned supine for 5 minutes prior to imaging to ensure fluid redistribution. A linear transducer (12 MHz) was used with neutral probe angle and minimal pressure. The anatomical landmark was the midpoint between the greater trochanter and the upper pole of the patella. Measurements included muscle thickness, pennation angle, fascicle length, echo intensity, cross-sectional area, and subcutaneous fat thickness. Images were taken in both transverse and longitudinal planes. Three measurements were taken per view to ensure accuracy.
Ultrasound Assessment of the Rectus Abdominis Muscle | At a single assessment visit
  The rectus abdominis muscle was assessed using the same ultrasound equipment and imaging protocol as for the rectus femoris. The anatomical reference point was located 3 cm lateral to the umbilicus, as per SARCUS group guidance. Images were acquired in both transverse and longitudinal planes. Measurements included muscle thickness, echo intensity, anatomical cross-sectional area, and subcutaneous fat thickness. Three measurements were taken per view to ensure reliability.

SECONDARY OUTCOMES:
Grip strength test | At a single assessment visit
  Accurate measurement of hand grip strength requires the use of a hand dynamometer (Jamar Plus) calibrated under well-defined (standardized) test conditions. Force values less than 16 Kg are considered positive.
Chair stand test | At a single assessment visit
  It can be used as an indicator of the strength of the lower limb muscles. It measures the amount of time a patient needs to get up five times from a sitting position without using their arms. It will help us to affirm that the person has a probable sarcopenia. Times greater than 15 seconds are considered positive.
Body Mass Index (BMI) | At a single assessment visit
  It is a measure used to assess a person's body weight in relation to their height. It is calculated by dividing a person's weight in kilograms by their height in meters squared (BMI = kg/m²).
Short Physical Performance Battery (SPPB) | At a single assessment visit
  Test to assess physical performance and degree of frailty consisting of 3 subtests: gait speed, balance, and lower limb strength. The maximum score is 12 points and a score ≤ 8 points indicates poor physical performance.
Gait speed | At a single assessment visit
  t is considered a fast, safe and very reliable test for sarcopenia, in a distance of 4 meters, values greater than 0.8 m/s are considered positive
Timed Up and Go (TUG) | At a single assessment visit
  A predictive test for frailty and falls, where individuals are asked to get up from a standard chair, walk to a marker 3 m away, turn around, and sit down again. Times greater than 20 seconds are considered positive.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Salamanca, Salamanca, Salamanca, Spain